CLINICAL TRIAL: NCT01395433
Title: A Single-dose, Open-label, Randomised, Crossover Bioequivalence Study in Healthy Young Men Comparing Two Formulations of Escitalopram
Brief Title: Bioequivalence Study Comparing Two Formulations of Escitalopram
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13154A; 2009-015108-24 (EudraCT Number)
Record Dates: First submitted 2011-07-13; First posted 2011-07-15 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: Assessing the bioequivalence of escitalopram dosage forms
MeSH Terms: interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Active Comparator): Conventional escitalopram
  Interventions: Drug: Escitalopram
- Treatment B (Experimental): Escitalopram test treatment B
  Interventions: Drug: Escitalopram
- Treatment C (Experimental): Escitalopram test treatment C
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — 2 x 10 mg, single dose
  Arms: Treatment A
Drug: Escitalopram — 2 x 10 mg, single dose
  Arms: Treatment B
Drug: Escitalopram — 1 x 20 mg, single dose
  Arms: Treatment C

SUMMARY:
This is a bioequivalence study, which is a regulatory requirement to ensure comparable in vivo performance, i.e. similarities in terms of safety and efficacy, after administration of two different dosage forms of escitalopram.

All subjects will receive three separate dosages of 20 mg escitalopram, which are 2 x 10 mg of the conventional dosage form (Treatment A) and 2 x 10 mg of the new dosage form being tested (Treatment B) and 1 x 20 mg of the new dosage form being tested (Treatment C). Test treatments B and C will each be compared to Treatment A, which is the active comparator (reference formulation).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 19 kg/m2 and 29 kg/m2, inclusive
* The subject is, in the opinion of the investigator, generally healthy based on assessment of medical history, physical examination, vital signs, electrocardiogram (ECG), and the results of the haematology, clinical chemistry, urinalysis, serology, and other laboratory tests

Exclusion Criteria:

* The subject has taken disallowed medication within 1 week prior to the first dose of investigational medicinal product (IMP), or within 5 half-lives prior to inclusion for any medication ingested, whichever is longer
* The subject has a significant history of drug or alcohol abuse
* The subject has taken any investigational products within 3 months prior to the first dose of IMP
* The subject has a history of or presence of any clinically significant immunological, cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, or psychiatric disease or other major disorder
* The subject has a history of cancer, other than basal cell or Stage 1 squamous cell carcinoma of the skin, which has not been in remission for at least 5 years prior to the first dose of IMP
* The subject has a history of abdominal surgery (excluding laparoscopic cholecystectomy or uncomplicated appendectomy) or thoracic or nonperipheral vascular surgery within 6 months prior to the first dose of IMP
* The subject has any concurrent illness that may affect the particular target or metabolism of the IMP
* The subject is, in the opinion of the investigator, unlikely to comply with the clinical study protocol or is unsuitable for any other reason

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To show bioequivalence on the basis of the area under the plasma concentration-time curve (AUC) and maximum observed plasma concentration (Cmax) of two different dosage forms of escitalopram | From the day of dosing up to 7 days in each dosing period
  The new dosage form being tested will be administered both as 2 x 10 mg and as 1 x 20 mg

SECONDARY OUTCOMES:
To investigate the safety and tolerability of the administration of the two dosage forms | Baseline + from the day of dosing up to 7 days in each dosing period
  Safety and tolerability parameters such as adverse advents, clinical safety laboratory tests and vital signs will be summarised using descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- NL001, Leiden, Netherlands

REFERENCES:
- [Result] Nilausen DO, Zuiker RG, van Gerven J. The perception and pharmacokinetics of a 20-mg dose of escitalopram orodispersible tablets in a relative bioavailability study in healthy men. Clin Ther. 2011 Oct;33(10):1492-502. doi: 10.1016/j.clinthera.2011.09.012. Epub 2011 Oct 13. PMID 21999886